CLINICAL TRIAL: NCT02887976
Title: An Open-label Extension (OLE), Expanded Access Study, to Assess Long-term Safety of SoluMatrix™ Abiraterone Acetate 500mg (4 x 125 mg qd) With Methylprednisolone (4mg Bid) in Patients Who Completed Study Number CHL-AA-201
Brief Title: Extension of SoluMatrix TM Abiraterone Acetate in Patients Who Completed Study Number CHL-AA-201
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GU Research Network, LLC (Other)
Collaborators: Churchill Pharmaceutical LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GURN-AA-201-OLE
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2016-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Castrate Resistant Prostate Cancer (CRPC); metastatic; castrate resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SoluMatrix™ Abiraterone Acetate (Experimental): SoluMatrix™ Abiraterone Acetate 500mg (4 x 125 mg qd) with Methylprednisolone (4mg bid)
  Interventions: Drug: SoluMatrix™ Abiraterone Acetate; Drug: Methylprednisolone

INTERVENTIONS:
Drug: SoluMatrix™ Abiraterone Acetate — SoluMatrix™ Abiraterone Acetate 500mg (4 x 125 mg qd) is an androgen synthesis inhibitor
  Other Names: Yonza
Drug: Methylprednisolone — Methylprednisolone (4mg bid) to maintain physiologic levels of corticosteroids which are reduced by SoluMatrix Abiraterone Acetate
  Other Names: medrol; solumedrol

SUMMARY:
An Open-label extension (OLE), expanded access study, to assess long-term safety of SoluMatrix™ Abiraterone Acetate 500mg (4 x 125 mg qd) with Methylprednisolone (4mg bid) in patients who completed study number CHL-AA-201.

DETAILED DESCRIPTION:
An Open-label extension (OLE), expanded access study, to assess long-term safety of SoluMatrix™ Abiraterone Acetate 500mg (4 x 125 mg qd) with Methylprednisolone (4mg bid) in patients who completed study number CHL-AA-201. An exploratory endpoint of Improved safety from switching from Zytiga (aberaterone Acetate 1000mg(4 x 250 mg qd) to SoluMatrix™ Abiraterone Acetate 500mg (4 x 125 mg qd) will also be ascertained..

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed
2. Previous, uninterrupted enrollment and treatment in trial number CHL-AA-201.

Exclusion Criteria:

1. Progressive disease as ascertained by the investigator using standard-of-care evaluations.
2. CHL-AA-201 D84 blood counts of the following:

   1. Absolute neutrophil count > 1500/µL
   2. Platelets > 100,000/µL
   3. Hemoglobin > 9 g/dL
3. CHL-AA-201 D84 chemistry values of the following:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x Upper Limit of Normal (ULN)
   2. Total bilirubin < 1.5 x ULN
   3. Creatinine< 1.5 x ULN
   4. Albumin > 3.0 g/dL
   5. Potassium > 3.5 mmol/L

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09; Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Month 9
  Safety as determined by adverse events deemed related to experimental treatment.

SECONDARY OUTCOMES:
Change in incidence of Treatment-Emergent Adverse Events in relation to Core Study | Month 9
  Explore if a reduction in adverse events occurs in subjects completing core study originally assigned to Zytiga Abiraterone Acetate plus prednison and switched to SoluMatrix Abiraterone Acetate plus methylprednisolone.,

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - GU Research Network/Wichita Urology Group, Wichita, Kansas
  - GU Research Network/Urology PC, Lincoln, Nebraska
  - GU Research Network/Urology Cancer Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
Peer reviewed Journal and/or professional meeting.